CLINICAL TRIAL: NCT07137598
Title: A Phase II, Multicenter, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of RO7790121 in Participants With Moderate to Severe Rheumatoid Arthritis Who Have an Inadequate Response or Intolerance to TNF and/or JAK Inhibitors
Brief Title: A Study to Assess the Efficacy and Safety of RO7790121 in Participants With Moderate to Severe Rheumatoid Arthritis Who Have Not Responded to or Who Cannot Tolerate Tumor Necrosis Factor (TNF) and/or Janus Kinase (JAK Inhibitors)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA45846
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Afimkibart Group I (Experimental): Participants will receive afimkibart via subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Afimkibart Group II (Experimental): Participants will receive afimkibart via SC injection.
  Interventions: Drug: Afimkibart
- Placebo (Placebo Comparator): Participants will receive afimkibart matched placebo via SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as SC injection.
  Other Names: PF 06480605; RVT-3101; RO7790121
  Arms: Afimkibart Group I; Afimkibart Group II
Drug: Placebo — Placebo will be administered as SC injection.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of Afimkibart (also known as RO7790121) compared with placebo in participants with moderate to severe rheumatoid arthritis (RA) who have an inadequate response or intolerance to TNF and/or JAK inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Has moderate to severe active RA defined by the presence of >=6 swollen joints and >=6 tender joints at screening and baseline (based on 66/68-joint count)
* Diagnosis of RA for >=3 months and also fulfills the 2010 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology (EULAR) classification criteria for RA
* Demonstrated an inadequate response or loss of response to or intolerance to >=1 conventional synthetic disease-modifying antirheumatic drug (csDMARD)

Exclusion Criteria:

* Have failed more than two TNF inhibitors or JAK inhibitors
* Class IV RA according to ACR revised response criteria (Hochberg et al. 1992)
* Past or current use of other biologic disease-modifying antirheumatic drugs (bDMARDs) (excluding TNF inhibitors) or rituximab
* Treatment with investigational therapy within 4 weeks or within 5 half-lives of the investigational therapy, whichever is longer, prior to initiation of study treatment.
* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA
* Has been treated with intra-articular, intramuscular, intravenous, trigger point or tender point, intra-bursa, or intra-tendon sheath corticosteroids in the preceding 8 weeks prior to the first dose of study drug
* History of a severe allergic reaction or anaphylactic reaction or known hypersensitivity to any component of the study drug (or its excipients) and/or other products in the same class
* Any major surgery within 6 weeks prior to screening or a major surgery planned during the study
* Any serious, chronic and/or unstable pre-existing medical, psychiatric, or other- condition
* History of malignancy, with the exception non-metastatic basal cell or cutaneous squamous cell cancer adequately treated with electrodesiccation and curettage or resection or in situ cervical cancer adequately treated and cured
* Participants with severe chronic or recurrent viral, bacterial, parasitic, or fungal infections
* History of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection
* History of organ transplant
* Any identified confirmed congenital or acquired immunodeficiency
* Abnormal laboratory values and liver function test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-04-17 (Estimated); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Disease Activity Score-28 for Rheumatoid Arthritis with C-Reactive Protein (DAS28-CRP) | Baseline, At Week 14

SECONDARY OUTCOMES:
Percentage of Participants Achieving an American College of Rheumatology 20 Percent (%), 50% or 70% Improvement (ACR20/ACR50/ACR70) | At Week 14
Change from Baseline Disease Activity Score-28 for Rheumatoid Arthritis with Erythrocyte Sedimentation Rate (DAS28-ESR) Score | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - Swollen Joint Count (SJC) | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - Tender Joint Count (TJC) | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS) | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - Patient's Global Assessment of Arthritis Pain-Visual Analog Scale (PGA Arthritis Pain-VAS) | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - Patient's Global Assessment of Disease Activity-Visual Analog Scale (PaGADA-VAS) | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - Health Assessment Questionnaire- Disability Index (HAQ-DI) | Baseline, At Week 14 and Week 24
Change From Baseline in the ACR Core Set - High-sensitivity C-reactive Protein (hsCRP) | Baseline, At Week 14 and Week 24
Change from Baseline in ACR20, ACR50 and ACR70 Response Rate | Baseline, At Week 24
Change from Baseline in Simplified Disease Activity Index (SDAI) Score | Baseline, At Week 14 and Week 24
Change from Baseline in Clinical Disease Activity Index (CDAI) Score | Baseline, At Week 14 and Week 24
Change from Baseline in Short Form-36 Health Survey (SF-36) Score | Baseline, At Week 14 and Week 24
Change from Baseline Disease Activity Score-28 for Rheumatoid Arthritis with C-Reactive Protein (DAS28-CRP) Score | Baseline, At Week 24
Percentage of Participants With Adverse Events (AEs) | Up to Week 38
Serum Concentration of RO7790121 at Specified Timepoints | Up to Week 38
Percentage of Participants With Anti-Drug Antibodies | Baseline, Up to Week 38

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (8):
  - SunValley Arthritis Center Ltd., Peoria, Arizona
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Accurate Clinical Research Inc., Lake Charles, Louisiana
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Accurate Clinical Management, Houston, Texas
  - DM Clinical Research, Tomball, Texas
  - Rheumatic Disease Center, Glendale, Wisconsin
- Bispebjerg og Frederiksberg Hospital, Frederiksberg, Denmark
- Hpital Cochin, Paris, Paris, France
- Poland (4):
  - Nzoz Bif-Med, Bytom
  - Centrum Kliniczno-Badawcze J. Brzezicki, B. Górnikiewicz-Brzezicka Lekarze Spó?ka Partne, Elbl?g
  - Zespol Poradni Specjalistycznych REUMED, Lublin
  - Reumatop Spolka Jawna, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing